CLINICAL TRIAL: NCT02704754
Title: Suvorexant and Trauma Related Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Howard University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GHUCCTS2015-1333
Record Dates: First submitted 2016-02-17; First posted 2016-03-10 (Estimated); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-01

CONDITIONS: Insomnia; Posttraumatic Stress Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- suvorexant (Experimental): 10mg administered before bedtime, during the first week; if well tolerated then the dose is increased to 20 mg before bedtime.
  Interventions: Drug: suvorexant
- Placebo pill (Placebo Comparator): A pill without active ingredients
  Randomization occurs 1:1 with stratification for gender and PTSD status.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: suvorexant — First in class orexin antagonist recently approved by the FDA for the treatment of insomnia
  Other Names: Belsomra
  Arms: suvorexant
Other: placebo — Pill with inactive ingredients
  Arms: Placebo pill

SUMMARY:
Problems sleeping are common after exposure to highly threatening experiences and can occur with and without a diagnosis of posttraumatic stress disorder (PTSD). Established treatments for PTSD are limited for addressing insomnia and many insomnia treatments appear to be limited in the context of PTSD. Suvorexant is FDA approved for insomnia and among approved drugs has a unique mechanism of action that may be well suited for targetting arousal at night dysregulated by trauma. The investigators will evaluate the efficacy of suvorexant for insomnia that developed in relation to trauma exposure, utilizing a placebo control, and polysomnography to identify biomarkers of response, in a six week trial.

DETAILED DESCRIPTION:
Disturbed sleep is one of the most common and distressing responses to exposure to severe trauma and can persist in many of those affected with and without accompanying posttraumatic stress disorder (PTSD). Insomnia is a risk factor for many of the conditions that are prevalent in trauma-exposed populations including PTSD, depression, and physical health conditions such as obesity, and cardiovascular disease. Trauma-related insomnia (TRI) is not typically differentiated in studies characterizing insomnia and its treatment, and insomnia accompanying PTSD has been shown to be relatively refractory to the treatments that are established for PTSD. Thus treatment of TRI presents an unmet need that has implications for the large and growing groups of people exposed to trauma in terms of relieving distress and preventing further psychiatric and medical morbidity.

Most of the data on TRI comes from research on populations with PTSD. Difficulty initiating and maintaining sleep is designated as one of the heightened arousal symptoms of PTSD in the DSM. Sleep studies have suggested increased wake after sleep onset (WASO), reduced slow wave sleep (SWS) in some PTSD populations and fragmented rapid eye movement (REM) sleep when PTSD is developing, and during its more acute stages. Suvorexant is a first in class orexin antagonist and is approved by the FDA for the indication of insomnia. Orexin antagonists dampen the activity of a specific arousal enhancing system in the brain during sleep. In rodent models suvorexant has been shown to enhance, and in healthy humans, to not affect slow wave and REM activity (in contrast with traditional hypnotics which can diminish both). Reducing arousal during sleep while reducing WASO and maintaining REM and slow wave sleep is a promising profile for the treatment of TRI. We are therefore proposing a placebo controlled evaluation to assess the efficacy of suvorexant for treating TRI with and without PTSD and its tolerability in these populations. We will include polysomnography (PSG) in order to have objective sleep outcomes and probe potential mechanisms and biomarkers predicting response. The proposed study will meet the objective below and test the following hypotheses:

Objective. To evaluate the efficacy of suvorexant for participants that meet criteria for insomnia and who identify a severely threatening event (DSM criterion A trauma) as a precipitant or a factor that significantly exacerbated their sleep disturbance.

The investigators hypothesize that suvorexant will improve subjective and objective indices of sleep disturbance; specifically, our primary outcome the polysomnographic (PSG) measure of sleep efficiency will be increased in the group receiving suvorexant compared with the group receiving placebo.

The effect of suvorexant versus placebo on the secondary outcome measures of the Insomnia Severity Index (ISI) scores and co-occurring symptoms of PTSD will also be evaluated.

Exploratory analyses will include comparison of response patterns among those with versus without significant symptoms of PTSD and relationships between increased in slow wave and rapid eye movement (REM) sleep and improvement in ISI scores and PTSD symptoms.

Adverse experiences and the tolerability of suvorexant in the recruited population with TRI will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy adults age 18-55 who meet DSM-5 criteria for insomnia and Criterion A (exposure to a traumatic event) for PTSD. The index trauma must have occurred within the past 5 years and at least 3 months before enrolling, and insomnia symptoms must have started or worsened after the exposure to the index trauma

Exclusion Criteria:

* Psychiatric disorders other than insomnia, PTSD and specific phobias; including bipolar and psychotic disorders and meeting criteria for DSM-5 moderate alcohol or drug use disorders within the past year.
* Diagnosis of a sleep disorder other than insomnia including PSG findings of apnea/hypopnea or periodic limb movement indices > 10/hour;
* Medical conditions that require consistent use of medication or compromise sleep;
* History of moderate to severe traumatic brain injury or mild traumatic brain injury with ongoing post-concussive symptoms;
* Suicidal ideation with intent to act or with specific plan and intent in the past 6 months (Type 4 - 5 ideation on the Columbia Suicide Severity Rating Scale) or a concerning history of prior suicidal behavior.
* Caffeine use exceeding 5 cups of coffee per day or its equivalent;
* Habitual bedtimes after 3 AM, habitual rise times after 10 AM, or habitual napping > 1hour/day;
* Pregnancy or breastfeeding, or expecting to conceive while in study;
* Positive urine toxicology.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Mellman, M.D., Principal Investigator — Howard University
Locations (1):
- Clinical Research Unit; Howard University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Reasonable requests will be accomodated via emailing the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: now, for 5 years
Access Criteria: reasonable request made directly to investigator

REFERENCES:
- [Background] Mellman TA, Birku K, Sandhu I, Lavela P, Kobayashi I. Evaluation of suvorexant for trauma-related insomnia. Sleep. 2022 May 12;45(5):zsac068. doi: 10.1093/sleep/zsac068. Epub 2022 Mar 18. PMID 35554590

RESULTS

PARTICIPANT FLOW:
Groups:
- Suvorexant: 10 to 20 mg to be administered before bedtime
  suvorexant: First in class orexin antagonist recently approved by the FDA for the treatment of insomnia
- Placebo Pill: A pill without active ingredients
  placebo: Pill with inactive ingredients
Period: Overall Study
Arm/Group | Suvorexant | Placebo Pill
Started | 21 | 20
Completed | 18 | 19
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant | Placebo Pill | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (12.7) | 35.4 (13.3) | 35.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 13 | 25
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37
Clinician Assessed PTSD Scale for DSM5 (CAPS-5) [Mean (Standard Deviation); unit: units on a scale] — Interview based on 0-4 severity of 20 items representing PTSD symptoms; total scale range 0 - 80, higher score is more severe.
  units on a scale | 8.8 (8.5) | 10.0 (7.1) | 9.38 (7.76)
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — 7 item scale, items 0-4, total score range 0 - 28, higher score indicates more severe insomnia
  units on a scale | 14.9 (4.7) | 16.6 (4.8) | 15.07 (4.03)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insomnia Severity Index Score From Baseline.
Description: A seven-item measure used to evaluate insomnia severity for the preceding two weeks. Items are scored on a 5-point scale and a total score ranging between 0 and 28 is obtained by summing the seven items, with higher scores indicating greater insomnia severity.
Time Frame: Baseline score minus 6 weeks or last observation (measure was also obtained at 2 and 4 weeks, the mathematical mean for the "last observation" was 5 weeks).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suvorexant | Placebo Pill
Number analyzed (Participants) | 18 | 19
units on a scale | 6.8 (5.0) | 8.6 (6.4)
Statistical Analysis 1: Comparison: Suvorexant vs Placebo Pill; Test type: Superiority; p < .05, t-test, 2 sided

2. Secondary Outcome: Change in Clinician Administered PTSD Scale Score
Description: Evaluates the frequency and intensity of each of the diagnostic symptoms of PTSD including nightmares and insomnia, total score was used which is a summation of all item scores, scores range between 0 to 80 with higher scores indicating more severe symptoms.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Suvorexant | Placebo Pill
Number analyzed (Participants) | 18 | 19
units on a scale | 4.2 (6.3) | 3.8 (5.2)

3. Secondary Outcome: Polysomnographically Measured Wake After Sleep Onset
Description: Polysomnography will provide objective measures of sleep, wake after sleep onset is the amount of wake time that occurs after initially falling asleep to the final awakening for the total sleep period measured in minutes.
Time Frame: Baseline values minus the values at 2 weeks.
Population: There were 5 patients in the suvorexant group and 6 in the placebo group who provided clinical ratings but for whom the second polysomnography was missed due to scheduling or was not scorable due to technical problems.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Suvorexant | Placebo Pill
Number analyzed (Participants) | 13 | 13
minutes | 21.0 (16.6) | 22.3 (11.6)

ADVERSE EVENTS:
Time Frame: Weeks 1, 2, 4, and 6 of medication treatment and 1-week following end of medication treatment
Arm/Group | Suvorexant | Placebo Pill
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 1/18 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suvorexant (N=18) | Placebo Pill (N=19)
sedation (Nervous system disorders) | 1 (1) | 0 (0) — moderate, remitted within 24 hours of last dose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT02704754/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT02704754/ICF_001.pdf